CLINICAL TRIAL: NCT00537680
Title: A Phase III Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy, Safety and Tolerability of Idebenone in the Treatment of Friedreich's Ataxia Patients
Brief Title: Study to Assess the Efficacy, Safety and Tolerability of Idebenone in the Treatment of Friedreich's Ataxia
Acronym: IONIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNT-III-002
Record Dates: First submitted 2007-09-07; First posted 2007-10-01 (Estimated); Results first posted 2011-12-29 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Friedreich's Ataxia
Keywords: Friedreich's Ataxia; Idebenone; ICARS
MeSH Terms: conditions — Friedreich Ataxia | interventions — idebenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 - 900 mg/day Idebenone (Experimental): mid dose Idebenone
  Interventions: Drug: Idebenone
- Arm 2 - up to 2250 mg/day Idebenone (Experimental): high dose Idebenone
  Interventions: Drug: Idebenone
- Arm 3 - Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Idebenone — Patients ≤ 45 kg/99 lbs: idebenone 450 mg/day; Patients > 45 kg/99 lbs: idebenone 900 mg/day
  Arms: Arm 1 - 900 mg/day Idebenone
Drug: Idebenone — Patients ≤ 45 kg/99 lbs: idebenone 1350 mg/day; Patients > 45 kg/99 lbs: idebenone 2250 mg/day
  Arms: Arm 2 - up to 2250 mg/day Idebenone
Drug: Placebo — Placebo was provided as film-coated tablets that were the same size, weight and appearance as the idebenone tablets.
  Arms: Arm 3 - Placebo

SUMMARY:
This study is meant to assess the effectiveness of idebenone on neurological outcome measures in patients with Friedreich's Ataxia over a 6 months period.

DETAILED DESCRIPTION:
The study involves 6 clinic visits and upon completion the possibility to join a 12 months extension study where all patients will receive high dose Idebenone.

ELIGIBILITY:
Inclusion criteria:

* Documented diagnosis of Friedreich's Ataxia (FRDA) with confirmed FRDA mutations
* Patients 8 - 17 years of age at baseline
* Patients with a body weight greater than 25 kg/55 lbs at baseline
* Patients able to walk at least 10 meters without accompanying person (ICARS Walking Capacities score ≤6) at screening and baseline
* Patients who in the opinion of the investigator are able to comply with the requirements of the study, including swallowing the study medication
* Negative urine pregnancy test at screening and baseline (female patients of childbearing potential)

Exclusion criteria:

* Treatment with idebenone, Coenzyme Q10 or vitamin E (if taken at a dose 5 times above the daily requirement) within the past month
* Patients with International Cooperative Ataxia Rating Scale (ICARS) score of greater than 54 or less than 10 at screening
* Pregnancy and/or breast-feeding
* Clinically significant abnormalities of clinical hematology or biochemistry including, but not limited to, elevations greater than 1.5 times the upper limit of normal of Aspartate Aminotransferase (AST; also known as GOT), Alanine Aminotransferase (ALT; also known as GPT) or creatinine
* History of abuse of drugs or alcohol
* Participation in the previous (Phase II) study of idebenone at the National Institutes of Health (NIH)
* Participation in a trial of another investigational drug within the last 3 months

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Perlman, MD, Principal Investigator — University of California, Los Angeles; David Lynch, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - David Geffen School of Medicine, UCLA, Los Angeles, California
  - The Children's Hopsital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Meier T, Perlman SL, Rummey C, Coppard NJ, Lynch DR. Assessment of neurological efficacy of idebenone in pediatric patients with Friedreich's ataxia: data from a 6-month controlled study followed by a 12-month open-label extension study. J Neurol. 2012 Feb;259(2):284-91. doi: 10.1007/s00415-011-6174-y. Epub 2011 Jul 22. PMID 21779958
- [Derived] Lagedrost SJ, Sutton MS, Cohen MS, Satou GM, Kaufman BD, Perlman SL, Rummey C, Meier T, Lynch DR. Idebenone in Friedreich ataxia cardiomyopathy-results from a 6-month phase III study (IONIA). Am Heart J. 2011 Mar;161(3):639-645.e1. doi: 10.1016/j.ahj.2010.10.038. Epub 2011 Jan 31. PMID 21392622
- [Derived] Lynch DR, Perlman SL, Meier T. A phase 3, double-blind, placebo-controlled trial of idebenone in friedreich ataxia. Arch Neurol. 2010 Aug;67(8):941-7. doi: 10.1001/archneurol.2010.168. PMID 20697044

RESULTS

PARTICIPANT FLOW:
Groups:
- Mid Dose Idebenone: 25 kg/55 lbs to ≤45 kg/99 lbs: idebenone 450 mg/day (1 x 150 mg tablet, t.i.d.) >45 kg/99 lbs: idebenone 900 mg/day (2 x 150 mg tablet, t.i.d.)
- High Dose Idebenone: 25 kg/55 lbs to ≤45 kg/99 lbs: idebenone 1350 mg/day (2 x 150 mg tablet, t.i.d.) >45 kg/99 lbs: idebenone 2250 mg/day (2 x 150 mg tablet, t.i.d.)
Period: Overall Study
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Started | 22 | 24 | 24
Completed | 22 | 22 | 24
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo | Total
Number analyzed (Participants) | 22 | 24 | 24 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 24 | 24 | 70
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.93 (2.54) | 13.44 (3.03) | 13.69 (2.77) | 13.68 (2.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 14 | 16 | 37
  Male | 15 | 10 | 8 | 33
Region of Enrollment [Number; unit: participants]
  United States | 22 | 24 | 24 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in the International Cooperative Ataxia Rating Scale (ICARS) From Baseline Assessment to Week 24
Description: International Cooperative Ataxia Rating Scale (ICARS):
  ICARS consists of a one-hundred-point semi-quantitative scale based upon 19 simple testing manoeuvres compartmentalized into postural and stance disorders, limb ataxia, dysarthria and oculomotor disorders and has been previously used in this patient population with good inter-rater reliability.
  Minimum score: 0, maximum score 100, higher score indicates greater impairment
  Calculation details: ICARS score at week 24 minus ICARS score baseline
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: ICARS points
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
ICARS points | -2.5 (6.3) | -2.4 (4.8) | -1.3 (4.4)

2. Secondary Outcome: Change in Friedreich's Ataxia Rating Scale (FARS) Scores From Baseline to Week 24
Description: To compare the efficacy of 6 months' treatment with 2 different doses of idebenone with that of placebo on neurological function as assessed by the Friedreich's Ataxia Rating Scale (FARS)
  FARS consists of a 25 manoeuvre exam along with 4 quantitative performance measures. The neurological exam covers bulbar function, upper limb coordination, lower limb coordination, peripheral nervous system function, deep tendon reflexes, stability and gait. The use of FARS has been recently validated as a sensitive scale for this population.
  The FARS exam scores can be added to make a total score ranging from 0 to 159. A higher score indicates a greater level of disability.
  Calculation details FARS score at week 24 minus FARS score baseline
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: FARS score
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
FARS score | -1.6 (6.52) | -1.2 (4.53) | 0.6 (5.91)

3. Secondary Outcome: Activities of Daily Living (ADL) of Friedreich's Ataxia Rating Scale (FARS), Change in ADL (Total Score ) From Baseline to Week 24
Description: To compare the efficacy of 6 months' treatment with 2 different doses of idebenone with that of placebo on Activities of Daily Living (ADL) assessed by the ADL scale of the Friedreich's Ataxia Rating Scale (FARS)
  score 0 to 36, higher score indicates greater impairment
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: ADL points
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
ADL points | 0.2 (2.45) | 0.6 (3.13) | 1.0 (2.97)

4. Secondary Outcome: Change in the International Cooperative Ataxia Rating Scale (ICARS) From Baseline Assessment to Week 12
Description: To compare the efficacy of 3 months' treatment with 2 different doses of idebenone with that of placebo on neurological impairment as assessed by the International Cooperative Ataxia Rating Scale (ICARS)
  International Cooperative Ataxia Rating Scale (ICARS):
  ICARS consists of a one-hundred-point semi-quantitative scale based upon 19 simple testing manoeuvres compartmentalized into postural and stance disorders, limb ataxia, dysarthria and oculomotor disorders and has been previously used in this patient population with good inter-rater reliability.
  Minimum score: 0, maximum score 100, higher score indicates greater impairment
  Calculation details: ICARS score at week 12 minus ICARS score baseline
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: ICARS points
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
ICARS points | -1.5 (5.35) | -1.6 (5.53) | -3.0 (3.52)

5. Secondary Outcome: Absolute Change From Baseline to Week 24 in the Relative Wall Thickness (RWT) of the Left Ventricle
Description: To compare the effects of idebenone on cardiac anatomy and function in patients with Friedreich's ataxia (FRDA) as assessed by echocardiography
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
cm | -0.032 (0.096) | 0.007 (0.071) | 0.010 (0.097)

6. Secondary Outcome: Percent Change From Baseline to Week 24 in the Relative Wall Thickness (RWT) of the Left Ventricle
Description: as for outcome 5
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
% change | -3.32 (15.300) | 1.53 (12.560) | 2.65 (17.135)

7. Secondary Outcome: Absolute Change From Baseline to Week 24 in Left Ventricular Mass Index (LVMI)
Description: as for outcome 5
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: g/m2
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
g/m2 | -3.06 (6.23) | -2.56 (4.27) | -1.26 (6.47)

8. Secondary Outcome: Percent Change From Baseline to Week 24 in Left Ventricular Mass Index
Description: as for outcome 5
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
% change | -4.5 (11.302) | -4.9 (8.713) | -1.7 (12.382)

9. Secondary Outcome: Absolute Change From Baseline to Week 24 in the Thickness of the Posterior Wall (PW) of the Left Ventricle
Description: as for outcome 5
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
cm | -0.018 (0.137) | -0.004 (0.112) | -0.038 (0.153)

10. Secondary Outcome: Percent Change From Baseline to Week 24 in the Thickness of the Posterior Wall (PW) of the Left Ventricle
Description: as for outcome 5
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
% change | -0.075 (13.379) | 0.12 (12.549) | -3.04 (14.651)

11. Secondary Outcome: Absolute Change From Baseline to Week 24 in the Thickness of the Interventricular Septum (IVS)
Description: as for outcome 5
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
cm | -0.014 (0.1983) | 0.021 (0.1474) | 0.063 (0.1952)

12. Secondary Outcome: Percent Change From Baseline to Week 24 in the Thickness of the Interventricular Septum (IVS)
Description: as for outcome 5
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Number analyzed (Participants) | 22 | 24 | 24
% change | 1.3 (18.160) | 2.6 (13.084) | 7.8 (19.480)

ADVERSE EVENTS:
Description: "0" means none.
Arm/Group | Mid Dose Idebenone | High Dose Idebenone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 2/24 | 0/24
Other Adverse Events (participants affected / at risk) | 18/22 | 23/24 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mid Dose Idebenone (N=22) | High Dose Idebenone (N=24) | Placebo (N=24)
idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mid Dose Idebenone (N=22) | High Dose Idebenone (N=24) | Placebo (N=24)
Infections (Infections and infestations) | 11 | 15 | 16
Nervous system disorders (Nervous system disorders) | 10 | 14 | 12
Gastrointestinal disorders (Gastrointestinal disorders) | 8 | 15 | 12
General disorders (General disorders) | 10 | 9 | 9
Musculoskeletal & connective tissue disorders (Musculoskeletal and connective tissue disorders) | 7 | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No